CLINICAL TRIAL: NCT03181516
Title: Efficacy and Safety of BB-12 Supplemented Strawberry Yogurt For Healthy Children on Antibiotics
Acronym: PLAY ON
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: Penn State University (Other); University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Daniel Merenstein, Professor and Director of Research Programs, Georgetown University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2016-1489
Record Dates: First submitted 2017-06-07; First posted 2017-06-08 (Actual); Results first posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Antibiotic-associated Diarrhea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BB-12 (Experimental): Bifidobacterium animalis subsp. lactis BB-12 (BB-12)-supplemented yogurt
  Interventions: Biological: Bifidobacterium animalis subsp. lactis BB-12
- Control (Placebo Comparator): Yogurt without Bifidobacterium animalis subsp. lactis BB-12
  Interventions: Other: Control

INTERVENTIONS:
Biological: Bifidobacterium animalis subsp. lactis BB-12 — Bifidobacterium animalis subsp. lactis BB-12-supplemented yogurt
  Arms: BB-12
Other: Control — Yogurt without Bifidobacterium animalis subsp. lactis BB-12
  Arms: Control

SUMMARY:
Probiotics are live microorganisms that, when administered in adequate amounts, confer a health benefit on the host. One of the most common indications for probiotic treatment is the prevention of antibiotic-associated diarrhea (AAD). Unfortunately, many probiotic products used for AAD are not supported by rigorous independent research, and often results in non-evidence-based usage. The overarching objective is to move research forward for the most well-studied Bifidobacterium strain. The primary aim is to test the efficacy of high dose, BB-12-supplemented yogurt in preventing AAD, compared to yogurt without BB-12, in children receiving antibiotics. Other aims are to further assess the safety of yogurt supplemented with BB-12, and to carry out longitudinal community structure and gene expression analysis of fecal microbiota to evaluate the impact of high dose BB-12 in a pediatric population receiving antibiotics. The microbiota includes hundreds of species, and its disruption is hypothesized to be an important factor in the development of AAD.

ELIGIBILITY:
Inclusion Criteria:

1. Child is between ages of 3-12 years
2. Caregiver has the ability to read, speak and write English or Spanish
3. Household has refrigerator for proper storage of drink
4. Household has telephone access
5. Enrollment must take place within 24 hours of starting antibiotics
6. Child was outpatient treated
7. Child was prescribed treatment with a penicillin or cephalosporin class antibiotic regimen for 7-10 days for a respiratory infection;

The following is a list (non-exhaustive) of inclusive antibiotics:

1. Amoxicillin
2. Augmentin (amoxicillin/clavulanate)
3. Ancef (cefazolin)
4. Cefadroxil
5. Cephalexin
6. Cephradine
7. Duricef (cefadroxil)
8. Keflex (cephalexin)
9. Kefzol (cefazolin)
10. Velosef (cephradine)
11. Ceclor (cefaclor)
12. Cefotan
13. Cefoxitin
14. Ceftin (cefuroxime)
15. Cefzil (cefprozil)
16. Lorabid (loracarbef)
17. Mefoxin (Cefoxitin)
18. Zinacef (cefuroxime)
19. Omnicef (cefdinir)
20. Suprax (cefixime)
21. Dicloxacillin
22. Pen-Vee K (penicillin)

Exclusion Criteria:

1. Developmental delays
2. Any chronic condition, such as diabetes or asthma, that requires medication
3. Prematurity, or born prior to 37 weeks gestation/of pregnancy
4. Congenital anomalies
5. Failure to thrive
6. Allergy to strawberry
7. Active diarrhea (diarrhea is defined in this study as three or more loose stools per day for two consecutive days)
8. Any other medicines used except anti-pyretic medicines (pro re nata concomitant medications are allowed)
9. Parental belief of lactose intolerance
10. History of heart disease, including valvulopathies or cardiac surgery, any implantable device or prosthetic
11. History of gastrointestinal surgery or disease
12. Milk-protein allergy
13. Allergy to any component of the product or the yogurt vehicle
14. Allergy or a hypersensitivity to the antibiotic prescribed by her/his provider
15. Allergy to any of the following medications:

    1. Tetracycline
    2. Erythromycin
    3. Trimethoprim
    4. Ciprofloxacin
16. blood oxygen saturation is less than 90% (if enrollment/baseline visit is completed in person and if the participant was prescribed antibiotics during a telemedicine visit)

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 255 (Actual)
Dates: Start 2017-09-30 (Actual); Primary Completion 2023-10-11 (Actual); Study Completion 2023-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Merenstein, MD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown University Department of Family Medicine, Research Division, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BB-12 | Control
Started | 125 | 130
Completed | 109 | 121
Not Completed | 16 | 9
Not completed — Withdrawal by Subject | 14 | 7
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BB-12 | Control | Total
Number analyzed (Participants) | 125 | 130 | 255
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Some participants did not fill out their birthday so their age was not known. However, it was confirmed that they were between the ages of 3-12 years old when enrolling.
  years
    number analyzed (Participants) | 110 | 113 | 223
    (all) | 6.97 (2.71) | 6.44 (2.87) | 6.70 (2.80)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: There were certain participants who did not answer the question regarding sex, so their sex was unknown causing the number of participants to differ.
  Participants
    number analyzed (Participants) | 118 | 126 | 244
    Female | 53 | 64 | 117
    Male | 65 | 62 | 127
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 58 | 58 | 116
  Not Hispanic or Latino | 61 | 68 | 129
  Unknown or Not Reported | 6 | 4 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 4 | 4 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 77 | 82 | 159
  More than one race | 19 | 17 | 36
  Unknown or Not Reported | 23 | 23 | 46
Region of Enrollment [Number; unit: participants]
  United States | 125 | 130 | 255
Health Insurance Status [Number; unit: participants]
  Yes | 110 | 123 | 233
  No | 10 | 4 | 14
  Unknown | 5 | 3 | 8
Smoking in the Household [Count of Participants; unit: Participants]
  Yes | 7 | 2 | 9
  No | 112 | 125 | 237
  Unknown | 6 | 3 | 9
Marital Status of Accompanying Guardian [Count of Participants; unit: Participants]
  Single | 16 | 12 | 28
  Married | 82 | 92 | 174
  Living with a Partner | 13 | 6 | 19
  Divorced | 4 | 2 | 6
  Separated | 2 | 5 | 7
  Widowed | 0 | 1 | 1
  Not reported/Unknown | 8 | 12 | 20
total annual income of all the family members living in the household before taxes [Count of Participants; unit: Participants]
  < $15,000 | 7 | 6 | 13
  $15,000 - $30,000 | 18 | 8 | 26
  $30,001 - $50,000 | 10 | 8 | 18
  $50,001 - $75,000 | 5 | 7 | 12
  $75,001 - $100,000 | 4 | 5 | 9
  $100,001 - $150,000 | 17 | 15 | 32
  $150,001 - $200,000 | 10 | 15 | 25
  > $200,000 | 29 | 29 | 58
  Prefer not to answer/Unknown | 25 | 37 | 62

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Diarrhea
Description: Diarrhea is clinically defined as three or more loose stools per day for two consecutive days. This will be a dichotomous (yes or no) outcome of diarrhea.
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | BB-12 | Control
Number analyzed (Participants) | 125 | 130
Participants
  Yes | 3 | 2
  No | 122 | 128

2. Primary Outcome: Adverse Events
Description: Number of reported adverse events over the duration of the study
Time Frame: Days 0-180
Measure: Number; unit: AE events
Arm/Group | BB-12 | Control
Number analyzed (Participants) | 125 | 130
AE events | 144 | 148

3. Secondary Outcome: Pediatric Quality-of-life Score
Description: The PedsQL Measurement Measurement Model for the Pediatric Quality-of-Life Inventory.
  Based on the PedsQL form filled out by participants, the scores were translated using the PedsQL form guidelines: 0=100, 1=75, 2=50,3=25,4=0. The raw scores of participants were averaged after translation. The lowest possible score is 0 and the highest possible score is 100. A higher score indicates a healthier lifestyle.
Time Frame: 7 days
Population: Some participants did not fill out the PEDSQL Day 7 form.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BB-12 | Control
Number analyzed (Participants) | 63 | 69
score on a scale | 85 (19) | 91 (10)

4. Secondary Outcome: Number of Events: Symptoms of Loose Stools, Constipation, Fever, Flatulence, Lack of Appetite, Pain, Rash, Vomiting, Cough, Earache, Nasal Congestion, Runny Nose, Sore Throat, Diarrhea.
Description: This will be a dichotomous (yes or no) outcome of loose stools, constipation, fever, flatulence, lack of appetite, pain, rash, vomiting, cough, earache, nasal congestion, runny nose, sore throat.
Time Frame: 14 days
Measure: Number; unit: Events
Arm/Group | BB-12 | Control
Number analyzed (Participants) | 125 | 130
Events
  Loose stools | 25 | 19
  Constipation | 15 | 21
  Fever | 11 | 14
  Flatulence | 6 | 4
  Lack of Appetite | 8 | 10
  Pain | 16 | 14
  Rash | 4 | 10
  Vomiting | 8 | 2
  Cough | 13 | 17
  Earache | 6 | 1
  Nasal Congestion | 14 | 12
  Runny nose | 10 | 9
  Sore throat | 5 | 13
  Diarrhea | 3 | 2

ADVERSE EVENTS:
Time Frame: 180 Days
Arm/Group | BB-12 | Control
All-Cause Mortality (participants affected / at risk) | 0/125 | 0/130
Serious Adverse Events (participants affected / at risk) | 0/125 | 0/130
Other Adverse Events (participants affected / at risk) | 64/125 | 69/130
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BB-12 (N=125) | Control (N=130)
Loose Stools (Gastrointestinal disorders) | 24 (25) | 17 (19)
Constipation (Gastrointestinal disorders) | 13 (15) | 18 (21)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (13) | 16 (17)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 13 (14) | 12 (12)
Fever (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 12 (14)
Pain (General disorders) | 16 (16) | 14 (14)
Runny Nose (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 9 (9)
Lack of Appetite (Gastrointestinal disorders) | 7 (8) | 10 (10)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 11 (13)
Rash (General disorders) | 4 (4) | 9 (10)
Flatulence (Gastrointestinal disorders) | 6 (6) | 3 (4)
Vomiting (General disorders) | 8 (8) | 2 (2)
Earache (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-28): https://cdn.clinicaltrials.gov/large-docs/16/NCT03181516/Prot_SAP_000.pdf